CLINICAL TRIAL: NCT04117568
Title: The Role of Emergency Neutrophils and Glycans in Postoperative and Septic Patients
Status: Terminated | Type: Observational
Why Stopped: Due to Covid-19 pandemic.
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Other Study IDs: AKB-Block
Record Dates: First submitted 2019-10-03; First posted 2019-10-07 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Sepsis; Septic Shock; Sepsis, Severe; Post-Op Complication; SIRS
MeSH Terms: conditions — Sepsis; Shock, Septic; Postoperative Complications | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood sampling — Blood sampling at 3-5 occasions per admission
  Other Names: No other intervention as this is an observational study

SUMMARY:
Surgical trauma elicits an immune response aiming to initiate healing and remove debris and damaged tissue locally at the wound site (1). This local reaction includes a considerable production of cytokines and chemokines that enters the circulation and initiate a systemic inflammatory response mediated by circulating cytokines and chemokines. This response is called systemic inflammatory immune response (SIRS) and is an aseptic systemic inflammation. Postoperative inflammation produces proinflammatory cytokines, mainly IL-6, IL1 beta, and tumor necrosis factor alfa (2). Neutrophils and emergency granulopoesis Polymorphonuclear neutrophils constitute the most abundant population of white blood cells. Their main task is to provide innate immune protection of the host from microbial attack, migrating to the site of infection, engulfing the microbes by phagocytosis, and killing the prey through attack by reactive oxygen species (ROS) and antimicrobial granule pro¬teins (22). Upon systemic infection or inflammation, e.g., sepsis or trauma, the bone marrow enters a state of emergency granulopoiesis, drenched in cytokines that augment production and survival of neutrophils for rapid delivery to the blood (23-25). Recently, advanced techniques have evolved that al¬low the isolation of different developmental stages of steady-state and emergency neutrophils, and characterization of these has just begun (26). Glycans Glycans (polysaccharides) attached to proteins and lipids on the surfaces on immune cells serve as ligands for glycan-binding proteins, lectins. Several neutrophil processes are directed by gly¬can - lectin interactions; selectin-directed rolling on the endothelium, siglec-mediated in¬hibitory signals, and activation of effector function by galectins. Many of the proteins that end up in neutrophil intra-cellular granules are highly glycosylated, but not much is known about if and how the neutrophil glycome evolves during the 'targeting-by-timing' process of differentiation and how this is affected by emergency granulopoiesis during systemic infection and inflammation. Here is a clear knowledge gap.

DETAILED DESCRIPTION:
Postoperative complications of any sort occurs in many of the patients undergoing high risk cancer surgery such as surgery for pancreatic, esophageal or ovarian malignancy (3, 4) These patients have a risk of wound infection mainly due to malnutrition and challenging surgical conditions (5, 6) A prolonged inflammatory response (overshoot) in some patients may lead to multiple organ failure (MOF) (7, 8).

Postoperative immunosuppression However, to handle the postoperative proinflammatory actions, patients also produce anti-inflammatory cytokines, mainly IL-4, IL-10 and IL-1 Ra. This is called compensatory inflammatory response syndrome (CARS). In cases of complications or malnutrition there may instead be an overshoot of the CARS mechanisms that lead to a suppression of the immune response (9, 10).

The surgical stress resulting in an imbalance in the inflammatory systems consume the circulating neutrophils and stresses the bone marrow to release immature, less efficient neutrophils, into the bloodstream, an event called emergency granulopoesis(11, 12).

Sepsis and ARDS Sepsis is one of the leading causes of death in Sweden and globally, and is characterized by an uncontrolled inflammatory reaction (13). The disease can affect everyone, including previously healthy people, and occurs when a normal bacterial infection invades the bloodstream and the body then responds with an inflammatory reaction. Acute organ dysfunction in sepsis primarily affects respiratory and circulatory systems (14). Pneumonia is the most common underlying cause of sepsis and respiratory insufficiency is the most common organ dysfunction in septic shock (15). Pneumonia with septic shock can develop into respiratory distress syndrome (ARDS) associated with a very high mortality rate, around 40% (16-18) Recently, ARDS was shown to be associated with migration of neutrophils, into the lung alveoli, and that such infiltration drives an inflammatory reaction, for which the pathophysiological mechanisms are incompletely mapped. Increased knowledge of the neutrophil role in ARDS could thus benefit the understanding of this complex syndrome(19, 20). In sepsis, the demand for enough circulating neutrophils to fight the infection is so high that reserve pools are exhausted and granulopoiesis switches to emergency mode. This results in release of immature neutrophils into circulation, the so-called left shift, used as an indicator of sepsis. As a result, circulating neutrophils in sepsis can be very heterogeneous, an effect also seen in autoimmune diseases and cancer (21). There are currently no tools to properly investigate these emergency neutrophil populations to utilize for diagnosis and disease follow-up.

Neutrophils and emergency granulopoesis Polymorphonuclear neutrophils constitute the most abundant population of white blood cells. Their main task is to provide innate immune protection of the host from microbial attack, migrating to the site of infection, engulfing the microbes by phagocytosis, and killing the prey through attack by reactive oxygen species (ROS) and antimicrobial granule pro¬teins (22). Upon systemic infection or inflammation, e.g., sepsis or trauma, the bone marrow enters a state of emergency granulopoiesis, drenched in cytokines that augment production and survival of neutrophils for rapid delivery to the blood (23-25). Recently, advanced techniques have evolved that al¬low the isolation of different developmental stages of steady-state and emergency neutrophils, and characterization of these has just begun (26). Glycans Glycans (polysaccharides) attached to proteins and lipids on the surfaces on immune cells serve as ligands for glycan-binding proteins, lectins. Several neutrophil processes are directed by gly¬can - lectin interactions; selectin-directed rolling on the endothelium, siglec-mediated in¬hibitory signals, and activation of effector function by galectins. Many of the proteins that end up in neutrophil intra-cellular granules are highly glycosylated, but not much is known about if and how the neutrophil glycome evolves during the 'targeting-by-timing' process of differentiation and how this is affected by emergency granulopoiesis during systemic infection and inflammation. Here is a clear knowledge gap.

Settings, research designs, patients and methods This project is a collaboration between the Sahlgrenska University Hospital, and Gothenburg University, Gothenburg, Sweden.

Adult patients (>18 years of age) are found from the surgical waiting list at the Sahlgrenska University hospital as they are assessed and scheduled for surgery for different kinds of malignancies, pancreatic malignancy, esophageal malignancy and ovarian malignancy. Furthermore, in a second study we will include patients undergoing cardiac surgery, with a heart lung machine in operation during the surgery. These patients will also be included from the surgical waiting list.

Patients in septic shock will be included from daily rounds at the central intensive care unit at the Sahlgrenska university Hospital. Septic shock is defined by criteria from Surviving sepsis campaign or sepsis III. As only around 30% of patients that are diagnosed with septic shock has a positive blood culture we will include both patients with or without a positive blood culture. After obtaining informed consent, patients will leave venous blood samples 3-5 times during their admission. The rationale for this was that we are not entirely sure of when patients may or may not enter the stage of emergency granulopoesis, but based on results from previous studies, and to achieve reasonable feasibility of the study protocol with as little missing data as possible these three sampling occasions seemed a reasonable compromise.

Clinical significance The basic characterization of glycome and glycoproteome in neutrophil granules will give in¬sights into, and be correlated with, the glycoconjugate status in the cell precursor populations that may be prematurely released from the bone marrow upon emergency granulopoiesis in¬duced by disease, such as sepsis, severe aseptic inflammation (trauma), autoimmune disease and cancer. Hence, our studies of neutrophils from blood and bone marrow, as well as emergency neutrophils from patients with sepsis and corresponding model systems will enable us not only to build mechanistic models and glycan databases, but also to develop novel diagnostic tools to identify and monitor disease. Here, our primary focus is sepsis and the subsequent development of ARDS. In ARDS neutrophils migrate into the alveoli of the lungs and degranulate in order to kill off bacteria. However, in the process lung tissue is injured and the inflammatory process causing severe hypoxemia and life threatening respiratory failure is fueled-on. As the glycome and glycoproteome seems to play a role in discriminating between harmful bacteria and endogenous structures it is of importance to clarify if there is any possible interactions that could be made to control this part of the destructive inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* undergoing surgery or presenting with sepsis according to definitions.

Exclusion Criteria:

* Interrupted surgery
* Neuropenia caused by cytostatics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postoperative patients or patients presenting with sepsis at Sahlgrenska University hospital, Gothenburg, Sweden
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Emergency granulopoesis in postoperative patients undergoing major surgery for malignancies. | 2019-2020
  Outcome : Is there an emergency granulopoesis in this category of patients? When does the granulopoesis occur? To what extent are the neutrophils affected by the emergency granulopoesis? Can the neutrophils produce reactive oxygen species?
Emergency granulopoesis perioperatively in patients undergoing cardiac surgery with the use of perioperative heart-lung machine. | 2020
  Is there an emergency granulopoesis in this category of patients? When does the granulopoesis occur? To what extent are the neutrophils affected by the emergency granulopoesis? Can the neutrophils produce reactive oxygen species?
Emergency granulopoesis in septic shock patients with and without a positive blood culture. | 2019-2020
  Is there an emergency granulopoesis in this category of patients? When does the granulopoesis occur? To what extent are the neutrophils affected by the emergency granulopoesis? Can the neutrophils produce reactive oxygen species?

CONTACTS AND LOCATIONS:
Overall Officials: Anna Karlsson-Bengtsson, Prof, Principal Investigator — Göteborg University
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No